CLINICAL TRIAL: NCT01014845
Title: A Phase 3, Randomized, Double-blind, Placebo (Hepatitis B Vaccine) Controlled Clinical Trial of Recombinant (E. Coli) Hepatitis E Vaccine
Brief Title: Clinical Trial of Recombinant Hepatitis E Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry); National Institute of Diagnostics and Vaccine Development in infectious disease (Unknown); Jiangsu Provincial Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro-HE-003; 2006AA02A209 (Other Grant/Funding Number: 863 Program of China)
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis E
Keywords: hepatitis E; vaccine; efficacy
MeSH Terms: conditions — Hepatitis E | interventions — hecolin; Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatitis E vaccine (Experimental): Hepatitis E vaccine, containing 30mcg of HEV239 recombinant antigen adsorbed to alum adjuvant suspended in 0.5ml phosphate buffer, was given at 0, 1, 6m for three doses.
  Interventions: Biological: hepatitis E vaccine
- HBV vaccine (Placebo Comparator): Hepatitis B vaccine, containing 5mcg of HBsAg recombinant antigen adsorbed to alum adjuvant suspended in 0.5ml phosphate buffer, was given at 0, 1, 6m for three doses.
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: hepatitis E vaccine — Intramuscularly given at 0, 1, 6m for three doses.
  Other Names: Hecolin
  Arms: Hepatitis E vaccine
Biological: Hepatitis B vaccine — Intramuscularly given at 0, 1, 6m for three doses.
  Arms: HBV vaccine

SUMMARY:
The primary purpose of this study is to determine whether the preventive hepatitis E are effective in the prevention of hepatitis E occurring at least 30 days after the administration of the third dose of vaccine.

The secondary purpose of this study is to to evaluate the safety and immunogenicity and immunopersistence of the study vaccine.

The initial study is planed to be ended on month 19 and the results were analysed and used for registration purpose. The extended study will be continued to assess the long-term efficacy, immunogenicity and safety.

DETAILED DESCRIPTION:
Participants were randomly allocated into two groups, one received Hepatitis E vaccine and the other received hepatitis B vaccine. The study was carried out with two stages. In the first stage (phase 3a), 2 645 subjects was enrolled and actively monitored for solicited adverse events for 1 month after each injection. Serum samples from all the subjects were collected on day 0, 7m, 13m, 19m and timely after then to evaluate the immunogenicity and immuno-persistency. In the second stage (phase 3b), another 109 959 subjects was enrolled and monitored for solicited adverse events for 1 month after each injection. Serum samples from 9764 subjects among the phase 3b participants were collected on day 0, 7m, 19m and timely after then to evaluate the immunogenicity and immuno-persistency. Serious adverse events during the trial were followed up.

Suspected hepatitis cases were identified through an established active hepatitis surveillance system. The sentinels of the system comprised all the healthcare facilities in the field. Suspected hepatitis was defined as when patients presented with systemic symptoms such as fatigue and/or loss of appetite for more than 3 days with alanine aminotransferase (ALT) exceeding 2.5 fold upper limit of normal range (ULN). Paired sera were obtained from these patients at the time of presentation and 2-6 weeks later. Sera were tested for the HEV antibodies and HEV-RNA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people aged from 16 years to 65 years old at the time of the first vaccination, normal intelligence and agree to sign the informed consent form.
* Subjects will reside in the study region in the next 19 months.
* Free of history of hepatitis B or hepatitis E.
* Can comply with the request of study.
* Axillary temperature is below 37 degree centigrade.

Exclusion Criteria:

For dose 1:

* Having other vaccine or immunoglobulin within two weeks;
* Having allergic history to vaccine and medicine
* Eclampsia, epilepsy, encephalopathy and history of mental disease or family;
* Thrombocytopenia or other disturbance of blood coagulation which would lead to muscle injection taboo;
* Fixed or suspected deficiency of immunologic function, containing immunosuppressant treatment(radiation therapy, chemical treatment, steroid hormone, antimetabolites, cytotoxic drugs), genetic defect(e.g. fabism), HIV or other factors;
* congenital malformation, eccyliosis or severe chronic disease(e.g. Down Syndrome, diabetes, sickle cell anemia or mental disease);
* fixed or suspected other disease including fever, active infection, liver and kidney disease, angiocardiopathy, malignancy, acute and chronic disease;
* joining other clinical study undergoing;
* women pregnant or in lactation.

For dose 2 or 3:

* Severe allergy for dose 1 or 2;
* Severe adverse reaction associated with last vaccination;
* New occurrence of symptoms meet dose 1 exclusion criteria after the first dose.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112604 (Actual)
Dates: Start 2007-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Rate of confirmed hepatitis E cases | One year since one month post the third injection

SECONDARY OUTCOMES:
IgG anti-HEV seroconversion rate | On one month post the third injection
Persistency of IgG anti-HEV | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, M.D., Study Director — National Institute of Diagnostics and Vaccine Development in infectious disease, Xiamen University; Feng-Cai Zhu, M.D., Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention, China
Locations (1):
- Dongtai Center for Disease Control and Prevention, Dongtai, Jiangsu, China

REFERENCES:
- [Background] Zhang J, Liu CB, Li RC, Li YM, Zheng YJ, Li YP, Luo D, Pan BB, Nong Y, Ge SX, Xiong JH, Shih JW, Ng MH, Xia NS. Randomized-controlled phase II clinical trial of a bacterially expressed recombinant hepatitis E vaccine. Vaccine. 2009 Mar 13;27(12):1869-74. doi: 10.1016/j.vaccine.2008.12.061. Epub 2009 Jan 23. PMID 19168109
- [Background] Li S, Tang X, Seetharaman J, Yang C, Gu Y, Zhang J, Du H, Shih JW, Hew CL, Sivaraman J, Xia N. Dimerization of hepatitis E virus capsid protein E2s domain is essential for virus-host interaction. PLoS Pathog. 2009 Aug;5(8):e1000537. doi: 10.1371/journal.ppat.1000537. Epub 2009 Aug 7. PMID 19662165
- [Background] He S, Miao J, Zheng Z, Wu T, Xie M, Tang M, Zhang J, Ng MH, Xia N. Putative receptor-binding sites of hepatitis E virus. J Gen Virol. 2008 Jan;89(Pt 1):245-249. doi: 10.1099/vir.0.83308-0. PMID 18089748
- [Background] Li SW, Zhang J, Li YM, Ou SH, Huang GY, He ZQ, Ge SX, Xian YL, Pang SQ, Ng MH, Xia NS. A bacterially expressed particulate hepatitis E vaccine: antigenicity, immunogenicity and protectivity on primates. Vaccine. 2005 Apr 22;23(22):2893-901. doi: 10.1016/j.vaccine.2004.11.064. PMID 15780738
- [Background] Zhang J, Gu Y, Ge SX, Li SW, He ZQ, Huang GY, Zhuang H, Ng MH, Xia NS. Analysis of hepatitis E virus neutralization sites using monoclonal antibodies directed against a virus capsid protein. Vaccine. 2005 Apr 22;23(22):2881-92. doi: 10.1016/j.vaccine.2004.11.065. PMID 15780737
- [Background] Li SW, Zhang J, He ZQ, Gu Y, Liu RS, Lin J, Chen YX, Ng MH, Xia NS. Mutational analysis of essential interactions involved in the assembly of hepatitis E virus capsid. J Biol Chem. 2005 Feb 4;280(5):3400-6. doi: 10.1074/jbc.M410361200. Epub 2004 Nov 22. PMID 15557331
- [Result] Zhu FC, Zhang J, Zhang XF, Zhou C, Wang ZZ, Huang SJ, Wang H, Yang CL, Jiang HM, Cai JP, Wang YJ, Ai X, Hu YM, Tang Q, Yao X, Yan Q, Xian YL, Wu T, Li YM, Miao J, Ng MH, Shih JW, Xia NS. Efficacy and safety of a recombinant hepatitis E vaccine in healthy adults: a large-scale, randomised, double-blind placebo-controlled, phase 3 trial. Lancet. 2010 Sep 11;376(9744):895-902. doi: 10.1016/S0140-6736(10)61030-6. Epub 2010 Aug 20. PMID 20728932
- [Result] Wu T, Huang SJ, Zhu FC, Zhang XF, Ai X, Yan Q, Wang ZZ, Yang CL, Jiang HM, Liu XH, Guo M, Du HL, Ng MH, Zhang J, Xia NS. Immunogenicity and safety of hepatitis E vaccine in healthy hepatitis B surface antigen positive adults. Hum Vaccin Immunother. 2013 Nov;9(11):2474-9. doi: 10.4161/hv.25814. Epub 2013 Jul 25. PMID 23887167
- [Result] Wu T, Zhu FC, Huang SJ, Zhang XF, Wang ZZ, Zhang J, Xia NS. Safety of the hepatitis E vaccine for pregnant women: a preliminary analysis. Hepatology. 2012 Jun;55(6):2038. doi: 10.1002/hep.25522. No abstract available. PMID 22161542
- [Result] Zhu FC, Huang SJ, Wu T, Zhang XF, Wang ZZ, Ai X, Yan Q, Yang CL, Cai JP, Jiang HM, Wang YJ, Ng MH, Zhang J, Xia NS. Epidemiology of zoonotic hepatitis E: a community-based surveillance study in a rural population in China. PLoS One. 2014 Jan 31;9(1):e87154. doi: 10.1371/journal.pone.0087154. eCollection 2014. PMID 24498033
- [Result] Zhang J, Zhang XF, Zhou C, Wang ZZ, Huang SJ, Yao X, Liang ZL, Wu T, Li JX, Yan Q, Yang CL, Jiang HM, Huang HJ, Xian YL, Shih JW, Ng MH, Li YM, Wang JZ, Zhu FC, Xia NS. Protection against hepatitis E virus infection by naturally acquired and vaccine-induced immunity. Clin Microbiol Infect. 2014 Jun;20(6):O397-405. doi: 10.1111/1469-0691.12419. Epub 2013 Nov 18. PMID 24118636
- [Derived] Huang S, Zhang X, Su Y, Zhuang C, Tang Z, Huang X, Chen Q, Zhu K, Hu X, Ying D, Liu X, Jiang H, Zang X, Wang Z, Yang C, Liu D, Wang Y, Tang Q, Shen W, Cao H, Pan H, Ge S, Huang Y, Wu T, Zheng Z, Zhu F, Zhang J, Xia N. Long-term efficacy of a recombinant hepatitis E vaccine in adults: 10-year results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2024 Mar 2;403(10429):813-823. doi: 10.1016/S0140-6736(23)02234-1. Epub 2024 Feb 19. PMID 38387470
- [Derived] Kmush BL, Yu H, Huang S, Zhang X, Wu T, Nelson KE, Labrique AB. Long-term Antibody Persistence After Hepatitis E Virus Infection and Vaccination in Dongtai, China. Open Forum Infect Dis. 2019 Mar 28;6(4):ofz144. doi: 10.1093/ofid/ofz144. eCollection 2019 Apr. PMID 31024978
- [Derived] Chen S, Zhou Z, Wei FX, Huang SJ, Tan Z, Fang Y, Zhu FC, Wu T, Zhang J, Xia NS. Modeling the long-term antibody response of a hepatitis E vaccine. Vaccine. 2015 Aug 7;33(33):4124-9. doi: 10.1016/j.vaccine.2015.06.050. Epub 2015 Jun 28. PMID 26126668
- [Derived] Zhang J, Zhang XF, Huang SJ, Wu T, Hu YM, Wang ZZ, Wang H, Jiang HM, Wang YJ, Yan Q, Guo M, Liu XH, Li JX, Yang CL, Tang Q, Jiang RJ, Pan HR, Li YM, Shih JW, Ng MH, Zhu FC, Xia NS. Long-term efficacy of a hepatitis E vaccine. N Engl J Med. 2015 Mar 5;372(10):914-22. doi: 10.1056/NEJMoa1406011. PMID 25738667